CLINICAL TRIAL: NCT00441896
Title: A Double-blind, Placebo-controlled, Dose-ranging Clinical Study to Evaluate the Safety, Tolerability, and Antiepileptic Activity of Ganaxolone in Treatment of Patients With Infantile Spasms
Brief Title: A Randomized, Controlled Trial of Ganaxolone in Patients With Infantile Spasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-0500
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Infantile Spasms
Keywords: infantile spasms; anticonvulsant; pediatric epilepsy; West Syndrome; epileptic spasms
MeSH Terms: conditions — Spasms, Infantile | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ganaxolone (Experimental): ganaxolone
  Interventions: Drug: Ganaxolone
- non-active drug (Placebo Comparator): placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ganaxolone
  Arms: ganaxolone
Other: Placebo
  Arms: non-active drug

SUMMARY:
The study consists of cohorts where participants are randomized, in a 2:1 ratio, to 1 of 2 sequences, A and B. In each cohort, Sequence A, comprised of participants, who will receive ascending doses of ganaxolone and ascending doses of placebo. Sequence B, comprised of participants, who will receive ascending doses of placebo and ascending doses of ganaxolone. The dosing level in each subsequent cohort will be based upon experience gained from previous cohorts.

DETAILED DESCRIPTION:
Male or female, 4 to 24 months of age (inclusive) with a diagnosis of IS with a 24 hour video EEG (vEEG) recording confirming the diagnosis and previously treated with 3 or fewer antiepileptic drugs (AEDs) are eligible for the study. The subject is able to continue treatment with concomitant AEDs (no more than 2; adrenocorticotropic hormone [ACTH], corticosteroids, felbamate, and vigabatrin are not allowed concomitantly). A ketogenic diet is permitted if it can be maintained for the duration of the study.

There will be a total of three weekly 24-hr video EEGs (baseline, end of weeks 1 and 2 of treatment). Dosing titration begins the day after each video EEG during the inpatient stay. All subjects will be receiving ganaxolone the day after the second video EEG.

A Data Monitoring Board (DMB) will determine whether successive cohorts of subjects can be dosed at an increased dose level; up to a maximum of 6 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with IS (regardless of etiology- except for a progressive neurologic illness). Diagnostic Criteria: Seizures consisting of single or repetitive short muscular contractions leading to flexion or extension. Spasms may be characterized as tonic or myoclonic contractions, may occur singly or in clusters, and typically occur bilaterally and symmetrically. The EEG pattern must be consistent with the diagnosis of IS (hypsarrhythmia, modified hypsarrhythmia, multifocal spike wave discharges, etc).
* Have a vEEG recording confirming the diagnosis of IS.
* Have had a magnetic resonance imaging (MRI) performed to determine any possible causes of IS.
* Have been previously treated with 3 or fewer AEDs.
* If being treated with concomitant AEDs

  * Current AEDs have been at a constant daily dose for at least 2 weeks; Note: Subjects with minor dose adjustments may be allowed to enter the study after shorter periods after detailed discussion with the medical monitor.
  * Have a stable clinical response/plateau for at least 2 weeks
  * Are able to continue treatment with no more than 2 concomitant AEDs (ACTH, corticosteroids, felbamate, and vigabatrin are not allowed concomitantly).
  * A ketogenic diet is permitted if it can be maintained for the duration of the study.
* Be a male or female, 4 to 24 months of age (inclusive)
* Have a Parent/Guardian who is properly informed of the nature and risks of the clinical study, who is willing and capable of complying with all clinical study procedures, and has given informed consent in writing prior to entering the clinical study
* Be able to participate for the full term of the clinical study.

Exclusion Criteria:

* Treatment with corticosteroids, ACTH, vigabatrin, felbamate, or any AED not approved by Regulatory Agencies, 2 weeks prior to randomization.
* Treatment with more than two AEDs at baseline.
* Have an active CNS infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive (with the exception of tuberous sclerosis) as evaluated by brain imaging (MRI).
* Have any disease or condition (medical or surgical) at screening that might compromise the hematologic, cardiovascular, pulmonary, renal, gastrointestinal, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the investigational product, or would place the subject at increased risk.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin greater than four times the upper limit of normal (ULN) or clinical laboratory value deemed clinically significant by the Investigator.
* History of recurrent status epilepticus.
* Have been exposed to any other investigational drug within 30 days prior to randomization.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, The Brain Institute, Miami, Florida
  - Child Neurology Care Center of Northwest Florida, Pensacola, Florida
  - Child Neurology Center of Northwest Florida, Pensacola, Florida
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - Montefiore Medical Center- Albert Einstein College of Medicine, The Bronx, New York
  - Le Bonheur Children's Medical Center, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: information about ganaxolone — https://marinuspharma.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, placebo-controlled, double-blind, dose-ranging study in which participants were randomized to ganaxolone:placebo in a 2:1 ratio into one of 5 cohorts. The primary focus of the study was to explore the dosing and titration schedule to help determine how rapidly infants can be titrated to a Maximum tolerated dose (MTD) to control spasms.
Groups:
- Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians 3 times a day (tid). Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 1 received starting doses of 3 milligrams per kilogram (mg/kg) tid with maximum allowable doses of 36 mg/kg/day (12 mg/kg tid).
- Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo: Participants were administered placebo followed by oral suspension of ganaxolone and then placebo using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 1 received starting doses of 3 mg/kg tid with maximum allowable doses of 36 mg/kg/day (12 mg/kg tid).
- Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 2 received starting doses of 6 mg/kg tid with maximum allowable doses of 45 mg/kg/day (15 mg/kg tid).
- Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo: Participants were administered placebo followed by oral suspension of ganaxolone and then placebo using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 2 received starting doses of 6 mg/kg tid with maximum allowable doses of 45 mg/kg/day (15 mg/kg tid).
- Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 3 received starting doses of 9 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
- Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo: Participants were administered placebo followed by oral suspension of ganaxolone and then placebo using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 3 received starting doses of 9 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
- Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 4 received starting doses of 12 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
- Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo: Participants were administered placebo followed by oral suspension of ganaxolone and then placebo using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 4 received starting doses of 12 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
- Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 5 received starting doses of 18 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
- Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo: Participants were administered placebo followed by oral suspension of ganaxolone and then placebo using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 5 received starting doses of 18 mg/kg tid with maximum allowable doses of 54 mg/kg/day (18 mg/kg tid).
Period: Overall Study
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Started | 6 | 3 | 7 | 4 | 12 | 3 | 7 | 5 | 6 | 4
Completed | 6 | 3 | 7 | 3 | 11 | 3 | 7 | 5 | 6 | 4
Not Completed | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received at least 1 dose of study medication
Groups:
- Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone: Participants were administered oral suspension of ganaxolone followed by placebo and then ganaxolone using an oral dosing syringe by hospital staff/parents/guardians tid. Each dose was separated by a minimum of 4 hours and a maximum of 8 hours. Participants in Cohort 1 received starting doses of 3 mg/kg tid with maximum allowable doses of 36 mg/kg/day (12 mg/kg tid).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo | Total
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 6 | 4 | 56
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.2 (2.48) | 20.3 (3.06) | 13.4 (4.89) | 23.0 (12.25) | 11.2 (5.47) | 14.0 (6.93) | 10.3 (4.96) | 13.2 (3.03) | 11.3 (3.27) | 11.5 (7.55) | 12.7 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 1 | 6 | 2 | 3 | 4 | 3 | 2 | 32
  Male | 3 | 0 | 2 | 3 | 5 | 1 | 4 | 1 | 3 | 2 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 9
  Not Hispanic or Latino | 5 | 3 | 5 | 4 | 10 | 1 | 5 | 4 | 6 | 4 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 2 | 0 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 9
  White | 3 | 2 | 7 | 1 | 6 | 3 | 5 | 3 | 1 | 3 | 34
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Frequency of Spasm Clusters at Day 10
Description: Spasm clusters were determined by a 24-hour video-electroencephalography (vEEG) at Day 10. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the Day 0 assessment before study drug infusion.
Time Frame: Baseline (Day 0) and Day 10
Population: Efficacy Population included all randomized participants who received at least 1 evaluation of efficacy at both Baseline (Day 0) and at either Visit 5 (Day 10) or Visit 8 (Day 20). Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Spasm clusters per day
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 5 | 3
Spasm clusters per day | 1.0 (20.06) | 2.7 (6.66) | -5.4 (10.97) | -1.0 (1.83) | -1.4 (13.69) | -5.3 (10.12) | -3.7 (4.92) | 0.2 (13.12) | -3.2 (5.02) | -1.7 (7.64)
Statistical Analysis 1: Comparison: Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.7391, ANCOVA
Statistical Analysis 2: Comparison: Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.5370, ANCOVA
Statistical Analysis 3: Comparison: Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.9080, ANCOVA
Statistical Analysis 4: Comparison: Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.2539, ANCOVA
Statistical Analysis 5: Comparison: Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.6657, ANCOVA

2. Secondary Outcome: Change From Baseline in Frequency of Spasm Clusters at Day 20
Description: Spasm clusters were determined by a 24-hour vEEG at Day 20. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the Day 0 assessment before study drug infusion.
Time Frame: Baseline (Day 0) and Day 20
Population: Efficacy Population.
Measure: Mean (Standard Deviation); unit: Spasm clusters per day
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 6 | 3
Spasm clusters per day | -3.2 (10.91) | 6.0 (11.53) | -5.0 (7.55) | -1.5 (3.11) | -1.1 (11.21) | -12.7 (26.27) | -4.4 (6.63) | -1.2 (13.85) | -3.2 (4.92) | -5.3 (7.57)
Statistical Analysis 1: Comparison: Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.4249, ANCOVA
Statistical Analysis 2: Comparison: Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.4177, ANCOVA
Statistical Analysis 3: Comparison: Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.3033, ANCOVA
Statistical Analysis 4: Comparison: Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.3014, ANCOVA
Statistical Analysis 5: Comparison: Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone vs Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo; Test type: Superiority; p = 0.1839, ANCOVA

3. Secondary Outcome: Number of Participants With Absence of Hypsarrhythmia
Description: Absence of hypsarrhythmia was determined by 24-hour vEEG at Day 10 and Day 20.
Time Frame: Day 10 and Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 6 | 3
Participants
  Day 10: number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 5 | 3
  Day 10 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 1 | 0
  Day 20 | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 2 | 3 | 0

4. Secondary Outcome: Number of Participants With Change in Clinical Status on the Investigator's Global Assessment
Description: The investigators rated the participants' overall clinical status based on 7 clinical factors: seizure frequency, duration, and intensity; adverse experiences; social, intellectual, and motor functioning. Using a 7-point scale ([1] marked improvement, [2] moderate improvement, [3] slight improvement, [4] no change from Baseline, [5] slight worsening, [6] moderate worsening, or [7] marked worsening). Higher score indicated worse symptoms. The investigators assessed the participants' status compared to their condition prior to initiating study medication.
Time Frame: Baseline (Day 0), Day 10 and Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 10 | 3 | 7 | 5 | 6 | 3
Participants
  Marked improvement at Day 10 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Moderate improvement at Day 10 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Slight improvement at Day 10 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 0
  No change from Baseline at Day 10 | 4 | 3 | 4 | 3 | 7 | 2 | 4 | 3 | 3 | 3
  Slight worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Marked improvement at Day 20 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Moderate improvement at Day 20 | 1 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1
  Slight improvement at Day 20 | 2 | 0 | 3 | 1 | 6 | 3 | 2 | 3 | 4 | 0
  No change from Baseline at Day 20 | 1 | 0 | 2 | 2 | 2 | 0 | 3 | 1 | 1 | 2
  Slight worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Moderate worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Change in Clinical Status on Caregiver's Global Assessment
Description: Caregiver global assessment of seizure severity and response to treatment rated the participants' based on 7 clinical factors: seizure frequency, duration, and intensity; adverse experiences; social, intellectual, and motor functioning. Using a 7-point scale ([1] marked improvement, [2] moderate improvement, [3] slight improvement, [4] no change from Baseline, [5] slight worsening, [6] moderate worsening, or [7] marked worsening). Higher score indicated worse symptoms. The assessment compared the participants' current status to their condition prior to initiating study medication.
Time Frame: Baseline (Day 0), Day10 and Day 20
Population: Efficacy population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 10 | 3 | 7 | 5 | 6 | 3
Participants
  Marked improvement at Day 10 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Moderate improvement at Day 10 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Slight improvement at Day 10 | 1 | 1 | 1 | 2 | 5 | 1 | 2 | 3 | 2 | 1
  No change from Baseline at Day 10 | 4 | 2 | 4 | 2 | 4 | 2 | 3 | 2 | 3 | 2
  Slight worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Moderate worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe worsening at Day 10 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Marked improvement at Day 20 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Moderate improvement at Day 20 | 1 | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 0
  Slight improvement at Day 20 | 2 | 0 | 2 | 1 | 6 | 2 | 3 | 3 | 4 | 0
  No change from Baseline at Day 20 | 1 | 0 | 3 | 2 | 2 | 0 | 2 | 0 | 1 | 3
  Slight worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Moderate worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe worsening at Day 20 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Spasm-free Durations
Description: Clinical spasms were determined by vEEG for at least 24 hours at Day 10 and Day 20. The number of participants with spasm-free duration have been presented.
Time Frame: Day 10 and Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 10 | 3 | 7 | 5 | 6 | 3
Participants
  Spasm-free Durations at Day 10 | 3 | 1 | 3 | 2 | 2 | 0 | 3 | 0 | 1 | 0
  Spasm-free Durations at Day 20 | 3 | 1 | 2 | 2 | 2 | 1 | 1 | 1 | 0 | 0

7. Secondary Outcome: Number of Participants With Seizure-free Days
Description: Seizure-free days were measured using data obtained from participants' daily dairy. Participants without seizures have been reported.
Time Frame: From Day 8 to Day 10 and From Day 18 to Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 10 | 3 | 7 | 5 | 6 | 3
Participants
  From Day 8 to Day 10 | 6 | 2 | 6 | 3 | 10 | 3 | 6 | 5 | 6 | 3
  From Day 18 to Day 20 | 6 | 1 | 6 | 4 | 10 | 3 | 6 | 5 | 6 | 3

8. Secondary Outcome: Number of Responders
Description: A responder is defined as a participant experiencing a greater than equal to (>=) 50 percent (%) decrease in spasm frequency. Test for responders was conducted by vEEG for up to 24 hours at Day 10 and Day 20
Time Frame: Day 10 and Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 6 | 3
Participants
  Day 10: number analyzed (Participants) | 6 | 3 | 7 | 4 | 11 | 3 | 7 | 5 | 5 | 3
  Day 10 | 2 | 1 | 3 | 0 | 3 | 0 | 2 | 2 | 2 | 1
  Day 20 | 2 | 0 | 4 | 2 | 3 | 1 | 4 | 1 | 1 | 1

9. Secondary Outcome: Developmental Assessment Using Denver-II Developmental Test at Day 20
Description: Denver-II Developmental Test measures a child's development in several areas:Personal-Social,Fine Motor-Adaptive,Language,and Gross Motor,from birth to 6 years old.It consists of 125 items that are organized into subscales and scored as pass,fail,or refused.To evaluate a child's progress,test compares their performance to a normative sample of children of same age.For each item,age at which 90% of children in normative sample pass it is determined.Derived score for each subscale is sum of item scores and represents difference between child's chronological age and age at which 90% of children in normative sample pass the items in that subscale.A higher derived score on a subscale indicates better performance on items in that subscale relative to other children of same age who have taken the test.Among subscales,Personal-Social subscale ranges from -16 months to 24 months;others range from - 12 months to 24 months.All subscales have a population mean of 0 and a standard deviation of 3.
Time Frame: At Day 20
Population: Efficacy Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
Number analyzed (Participants) | 5 | 3 | 7 | 3 | 11 | 2 | 7 | 5 | 5 | 3
Scores on a scale
  Personal Social at Day 20 | -5.48 (1.618) | -16.90 (2.563) | -8.79 (5.874) | -8.73 (6.071) | -7.76 (3.727) | -5.35 (0.354) | -5.99 (4.354) | -10.22 (4.925) | -7.72 (4.581) | -12.93 (7.336)
  Fine Motor Adaptive at Day 20 | -4.38 (1.834) | -14.63 (2.409) | -7.49 (5.414) | -7.70 (5.624) | -6.40 (4.224) | -5.05 (2.051) | -6.16 (4.484) | -10.24 (6.080) | -8.32 (3.637) | -12.87 (7.731)
  Language at Day 20 | -1.36 (2.681) | -12.33 (4.196) | -7.23 (7.020) | -5.17 (3.017) | -5.82 (3.880) | -4.95 (0.778) | -6.09 (4.674) | -8.22 (5.644) | -7.44 (3.089) | -10.77 (7.223)
  Gross Motor at Day 20 | -3.96 (2.532) | -13.63 (2.079) | -7.16 (5.298) | -7.00 (5.828) | -5.58 (3.329) | -3.00 (2.546) | -6.89 (4.282) | -8.74 (5.546) | -8.76 (3.260) | -13.43 (8.618)

ADVERSE EVENTS:
Time Frame: Up to 25 days
Description: AEs and SAEs were collected in ITT Population, which included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3 | 0/7 | 0/4 | 0/11 | 0/3 | 0/7 | 0/5 | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 0/7 | 0/4 | 0/11 | 0/3 | 2/7 | 0/5 | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 5/7 | 1/4 | 9/11 | 1/3 | 4/7 | 2/5 | 4/6 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=6) | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo (N=3) | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=7) | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo (N=4) | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=11) | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo (N=3) | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=7) | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo (N=5) | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=6) | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo (N=4)
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=6) | Cohort 1: Sequence B: Placebo/Ganaxolone/Placebo (N=3) | Cohort 2: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=7) | Cohort 2: Sequence B: Placebo/Ganaxolone/Placebo (N=4) | Cohort 3: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=11) | Cohort 3: Sequence B: Placebo/Ganaxolone/Placebo (N=3) | Cohort 4: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=7) | Cohort 4: Sequence B: Placebo/Ganaxolone/Placebo (N=5) | Cohort 5: Sequence A: Ganaxolone/Placebo/Ganaxolone (N=6) | Cohort 5: Sequence B: Placebo/Ganaxolone/Placebo (N=4)
Somnolence (Nervous system disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Puncture site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Teething (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pityriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spitting up (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No